CLINICAL TRIAL: NCT06983795
Title: Pioneering Advancements in Cardiocerebrovascular Interactions in the Asia pacFIC - Patent Foramen Ovale Study
Acronym: PACIFIC-PFO
Status: Not yet recruiting | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: PACIFIC-PFO
Record Dates: First submitted 2025-02-28; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-10

CONDITIONS: Ischemic Stroke; Patent Foramen Ovale
Keywords: Patent Foramen Ovale; Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke; Foramen Ovale, Patent | interventions — Practice Management, Medical; Clopidogrel; Ticagrelor; Dipyridamole; Cilostazol; N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients diagnosed with patient foramen ovale and ischemic stroke or transient ischemic attack.: The PACIFIC-PFO registry aims to include patients from Asia and Oceania. Academic, non-academic, urban and rural sites will be included. Principal investigators will be neurologists or cardiologists. A confirmed diagnosis of ischemic stroke or TIA is mandatory before enrolment. Information on the interventions performed and treatment instigated (e.g. PFO closure, medical therapy) will be collected.
  Interventions: Procedure: PFO closure using approved PFO closure devices, Surgical PFO closure; Drug: Medical management

INTERVENTIONS:
Procedure: PFO closure using approved PFO closure devices, Surgical PFO closure — PFO closure using approved PFO closure devices, Surgical PFO closure
  Other Names: Amplatzer™ Septal Occluder; Amplatzer™ PFO Occluder; Amplatzer™ Cribriform (for a septum with more than one hole); Gore® Cardioform Septal Occluder; Gore® Cardioform ASD Occluder (for larger ASDs); STARFlex® Septal Closure System
Drug: Medical management — Antiplatelet therapy
  * ASA, also called acetylsalicylic acid (Aspirin, Asaphen, Entrophen, Novasen)
  * clopidogrel (Plavix)
  * ticagrelor (Brilinta)
  * dipyridamole (Persantine)
  * cilostazol
  Anticoagulation therapy
  * apixaban (Eliquis)
  * dabigatran (Pradaxa)
  * edoxaban (Lixiana)
  * rivaroxaban (Xarelto)
  * warfarin (Coumadin)
  Other Names: Antiplatelet therapy e.g. aspirin, clopidogrel, ticagrelor, dipyridamole, cilostazol, or a combination of these medications; Anticoagulation e.g warfarin, direct oral anticoagulants

SUMMARY:
A registry of patients from the Asia-Pacific region with PFO and ischemic stroke, designed to study the characteristics, investigations, treatment and outcomes using real-world data.

DETAILED DESCRIPTION:
This is an observational, multi-center, non-randomized real-world registry including ischemic stroke and/or transient ischemic attack patients with PFO in the Asia Pacific region. The primary objective of this registry is to assess the clinical characteristics and outcomes of patients with PFO and stroke or TIA using real-world data in the Asia-Pacific region, including patients who underwent PFO closure versus medical management only.

Patients who had ischemic stroke or TIA within 5 years of inclusion into the registry, with follow up data of at least 1 year. Patients with AIS or TIA within one year of inclusion into the registry will be part of the prospective cohort. The total duration of the registry will be approximately 3 years.

ELIGIBILITY:
Inclusion Criteria

1. Subject has experienced acute ischemic stroke or transient ischemic attack
2. Subject is screened with presence of PFO (right-to-left shunt) on appropriate cardiac imaging (transthoracic echocardiography and/or transesophageal echocardiography) or transcranial Doppler bubble study
3. Age ≥18 years

Exclusion Criteria

1. Stroke mimics, haemorrhagic stroke or cerebral venous thrombosis
2. Subjects with less than 3 months of follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke or TIA and PFO identified would be screened for inclusion into the PACIFIC-PFO registry. Consecutive patients should be identified for inclusion by the local research team in each participating centers. Reason for exclusion after screening should be clearly stated and documented on a Screening and Enrollment Log, in order to minimize bias.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Recurrent ischemic stroke or transient ischemic attack event within 1 year | Within 1 year
  Ischemic stroke is defined as:
  Acute focal neurological dysfunction caused by focal infarction at single or multiple sites of the brain or retina. Evidence of acute infarction may come either from A) Symptom duration lasting more than 24 hours B) Neuroimaging or other technique in the clinically relevant area of the brain
  TIA is defined as:
  A transient episode of focal neurological dysfunction caused by focal brain or retinal ischemia without acute infarction in the clinically relevant area of the brain or retina.
  Symptoms should resolve completely within 24 hours.

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) | 90 days
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6, running from perfect health without symptoms to death.
Short term and long term neurological and cardiovascular outcomes | 90 days, 1 year, >1 year
  1. Recurrent stroke or TIA
  2. Systemic embolism
  3. Acute myocardial infarction
  4. Cardiovascular mortality
  5. All-cause mortality
  6. Major and minor bleeding defined according to the ISTH criteria
  7. Intracranial hemorrhage

OTHER OUTCOMES:
To validate PFO risk stratification scores in an Asia-Pacific cohort - RoPE score | 5 years
  PFO risk stratification scores are widely used to determine the likelihood that PFO discovered in the setting of an otherwise-cryptogenic stroke was pathogenically related to the stroke rather than an incidental finding.
  ROPE score The RoPE score ranges from 0 to 10, with scores of 0 to 3 indicating a negligible likelihood that the stroke is attributable to the PFO and a score of 10 indicating an approximately 90% probability that the stroke is attributable to the PFO.
To validate PFO risk stratification scores in an Asia-Pacific cohort - PASCAL score | 5 years
  PFO risk stratification scores are widely used to determine the likelihood that PFO discovered in the setting of an otherwise-cryptogenic stroke was pathogenically related to the stroke rather than an incidental finding.
  PASCAL score PASCAL combines the RoPE score with the presence or absence of high-risk PFO features to determine the likelihood that the PFO was causally related to the index stroke
To validate PFO risk stratification scores in an Asia-Pacific cohort - Spencer Grading | 5 years
  PFO risk stratification scores are widely used to determine the likelihood that PFO discovered in the setting of an otherwise-cryptogenic stroke was pathogenically related to the stroke rather than an incidental finding.
  Spencer algorithm grading scale with transcranial Doppler bubble study methodology
To evaluate the impact of access to PFO closure and availability of heart-brain teams on patient outcomes | 5 years
  The outcomes of the patients will be compared between centres with PFO closures services and heart-brain teams with those without. Patients treated by a heart-brain multi-disciplinary team were compared to those who were not.
To compare our regional data with other real-world registries or clinical trial data | 5 years
  To compare the patient characteristics, investigations, treatment and management in this regional registry with other published registries or clinical trials.
Other objectives | 5 years
  To identify other variables associated with PFO-related stroke specific to the Asian population, and to develop Asian-specific risk stratification methods which may have higher predictive values. Exploratory analysis of patients with PFO closure will be performed, for outcomes such as incidence of atrial fibrillation.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to restrictions stipulated by Ethics Approval.

REFERENCES:
- [Background] Saver JL, Mattle HP, Thaler D. Patent Foramen Ovale Closure Versus Medical Therapy for Cryptogenic Ischemic Stroke: A Topical Review. Stroke. 2018 Jun;49(6):1541-1548. doi: 10.1161/STROKEAHA.117.018153. Epub 2018 May 14. No abstract available. PMID 29760277
- [Background] Kim JS, Thijs V, Yudi M, Toyoda K, Shiozawa M, Zening J, Clapp B, Albers B, Diener HC. Establishment of the Heart and Brain Team for Patent Foramen Ovale Closure in Stroke Patients: An Expert Opinion. J Stroke. 2022 Sep;24(3):345-351. doi: 10.5853/jos.2022.02103. Epub 2022 Sep 30. PMID 36221937
- [Background] Toh KZX, Koh MY, Ho JSY, Ong KHX, Lee YQ, Chen X, Fang JT, Chong EY, Lim ICZY, Teo YH, Teo YN, Chua CYK, Lim Y, Chan BPL, Sharma VK, Yeo LLL, Sia CH, Tan BYQ. Potential Embolic Sources in Embolic Stroke of Undetermined Source Patients with Patent Foramen Ovale. Cerebrovasc Dis. 2023;52(5):503-510. doi: 10.1159/000527791. Epub 2022 Dec 1. PMID 36455524
- [Background] Diener HC, Akagi T, Durongpisitkul K, Thomson VS, Prabhakar AT, Sharpe R, Albers B, Lewalter T, Oki K, Sharma VK. Closure of the patent foramen ovale in patients with embolic stroke of undetermined source: A clinical expert opinion and consensus statement for the Asian-Pacific region. Int J Stroke. 2020 Dec;15(9):937-944. doi: 10.1177/1747493020941658. Epub 2020 Jul 17. PMID 32677579
- [Background] Kent DM, Saver JL, Ruthazer R, Furlan AJ, Reisman M, Carroll JD, Smalling RW, Juni P, Mattle HP, Meier B, Thaler DE. Risk of Paradoxical Embolism (RoPE)-Estimated Attributable Fraction Correlates With the Benefit of Patent Foramen Ovale Closure: An Analysis of 3 Trials. Stroke. 2020 Oct;51(10):3119-3123. doi: 10.1161/STROKEAHA.120.029350. Epub 2020 Sep 14. PMID 32921262
- [Background] Kent DM, Saver JL, Kasner SE, Nelson J, Carroll JD, Chatellier G, Derumeaux G, Furlan AJ, Herrmann HC, Juni P, Kim JS, Koethe B, Lee PH, Lefebvre B, Mattle HP, Meier B, Reisman M, Smalling RW, Soendergaard L, Song JK, Mas JL, Thaler DE. Heterogeneity of Treatment Effects in an Analysis of Pooled Individual Patient Data From Randomized Trials of Device Closure of Patent Foramen Ovale After Stroke. JAMA. 2021 Dec 14;326(22):2277-2286. doi: 10.1001/jama.2021.20956. PMID 34905030
- [Background] Kent DM, Ruthazer R, Weimar C, Mas JL, Serena J, Homma S, Di Angelantonio E, Di Tullio MR, Lutz JS, Elkind MS, Griffith J, Jaigobin C, Mattle HP, Michel P, Mono ML, Nedeltchev K, Papetti F, Thaler DE. An index to identify stroke-related vs incidental patent foramen ovale in cryptogenic stroke. Neurology. 2013 Aug 13;81(7):619-25. doi: 10.1212/WNL.0b013e3182a08d59. Epub 2013 Jul 17. PMID 23864310
- [Background] Turc G, Calvet D, Guerin P, Sroussi M, Chatellier G, Mas JL; CLOSE Investigators. Closure, Anticoagulation, or Antiplatelet Therapy for Cryptogenic Stroke With Patent Foramen Ovale: Systematic Review of Randomized Trials, Sequential Meta-Analysis, and New Insights From the CLOSE Study. J Am Heart Assoc. 2018 Jun 17;7(12):e008356. doi: 10.1161/JAHA.117.008356. PMID 29910193
- [Background] Overell JR, Bone I, Lees KR. Interatrial septal abnormalities and stroke: a meta-analysis of case-control studies. Neurology. 2000 Oct 24;55(8):1172-9. doi: 10.1212/wnl.55.8.1172. PMID 11071496
- [Background] Koutroulou I, Tsivgoulis G, Tsalikakis D, Karacostas D, Grigoriadis N, Karapanayiotides T. Epidemiology of Patent Foramen Ovale in General Population and in Stroke Patients: A Narrative Review. Front Neurol. 2020 Apr 28;11:281. doi: 10.3389/fneur.2020.00281. eCollection 2020. PMID 32411074